CLINICAL TRIAL: NCT07128121
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Immunogenicity of the Respiratory Syncytial Virus IN006 Bivalent mRNA Vaccine (IN006) in Healthy Participants Aged 60 Years and Older
Brief Title: A Phase 2 Study to Describe the Safety and Immunogenicity of Respiratory Syncytial Virus Vaccine IN006 in Healthy Participants Aged 60 Years and Older
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen Shenxin Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IN006003
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Syncytial Virus (RSV) Infection
Keywords: mRNA Vaccine; IN006; Respiratory syncytial virus; RSV; Viral Diseases; Messenger RNA; Innorna; Shenxin; Vaccines; Respiratory tract infections; Safety; Reactogenicity; Immunogenicity
MeSH Terms: conditions — Infections; Virus Diseases; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IN006 Dose A (Arm 1) (Experimental): One injection of Dose A of IN006 on Day 0. Participants will be further randomized to receive a second injection of either IN006 at Dose A or matching-placebo approximately 12 months later. Participants receive a second injection of placebo will be further randomized to receive a third injection of either IN006 at Dose A or matching-placebo approximately 24 months later.
  Interventions: Biological: Respiratory Syncytial Virus IN006 Bivalent mRNA Vaccine (IN006)
- IN006 Dose B (Arm 2) (Experimental): One injection of Dose B of IN006 on Day 0. Participants will be further randomized to receive a second injection of either IN006 at Dose B or matching-placebo approximately 12 months later. Participants receive a second injection of placebo will be further randomized to receive a third injection of either IN006 at Dose B or matching-placebo approximately 24 months later.
  Interventions: Biological: Respiratory Syncytial Virus IN006 Bivalent mRNA Vaccine (IN006)
- Placebo (Arm 3) (Placebo Comparator): Placebo On injection of placebo on Day 0.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Respiratory Syncytial Virus IN006 Bivalent mRNA Vaccine (IN006) — Formulation for injection
  Arms: IN006 Dose A (Arm 1); IN006 Dose B (Arm 2)
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo (Arm 3)

SUMMARY:
The study will evaluate the safety, tolerability, and immunogenicity of 2 dose levels of IN006 in healthy participants who aged at 60 years or older; of a revaccination of IN006 given 12 months or 24 months after the initial vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants aged ≥60 years, male or female.
2. The participants signed the informed consent form, and were able to provide valid identification documents. They also understood and complied with the requirements of the trial protocol.
3. Female participants must be non-childbearing potential. If male participants have female partners of childbearing potential, they must agree to use effective contraception from the signing of informed consent until 6 months after each vaccination.
4. Participants must be capable of performing self-care and routine activities of daily living.

Exclusion Criteria:

1. Body Mass Index (BMI) <18 kg/m^2 or ≥30 kg/m^2.
2. During the screening period, laboratory test results were abnormal and had clinical significance, or the severity reached or exceeded the Grade 2 criteria; or 12-lead electrocardiogram results were abnormal and had clinical significance (except for heart rate, for which the criterion relevant to pulse rate in exclusion criterion #3 should be applied). (For laboratory tests, a retest can be conducted at the discretion of investigators to determine the eligibility of the participants).
3. Vital signs meeting any of the following:

   * Systolic blood pressure <90 mmHg and/or diastolic blood pressure <50 mmHg;
   * Poorly controlled hypertension: systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg;
   * Pulse rate >100 beats per minute or <50 beats per minute;
   * Axillary temperature >37.0°C.
4. Tattoos, scars, bruises, or other conditions at the injection site that may interfere with local reaction assessment.
5. Known allergy to the investigational vaccine or its excipients, or history of severe allergic reactions to other vaccines, foods, or medications.
6. Previously received any investigational or licensed Respiratory Syncytial Virus (RSV) vaccine, or administration of investigational/licensed RSV prophylactic monoclonal antibodies within the last 6 months.
7. Received inactivated, subunit, or recombinant influenza vaccine within 14 days prior to randomization, or any other vaccine within 28 days prior to randomization; Or plan to receive any vaccines within 28 days after the investigational vaccine.
8. Use of antipyretics, analgesics, or anti-allergic drugs within 3 days prior to randomization.
9. Have received blood or blood-related products (including immunoglobulins) within 3 months prior to randomization, or had planned to use during the trial.
10. Participants with the following diseases (based on inquiry and/or relevant diagnosis):

    * A history of acute respiratory infection within 2 weeks of randomization; Or a history of confirmed RSV-associated respiratory infection within 3 months prior to vaccination; Or during the screening, RSV IgM is positive;
    * Any acute illness or acute exacerbation of a chronic illness within 3 days prior to randomization;
    * History of congenital or acquired immune deficiency or autoimmune diseases, or long-term use (continuous use > 14 days) of corticosteroids (dose ≥ 20mg/day prednisone or equivalent dose) or other immunosuppressants within the past 6 months;
    * Participants who have been diagnosed with or currently have an infectious disease (including hepatitis B, hepatitis C, and acquired immune deficiency syndrome), those who currently have active tuberculosis, or those whose tests for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus antibody are positive;
    * Previous or current neurological disorders (excluding seizures other than febrile seizures in children, and other types of epilepsy); History or family history of mental illness;
    * Asplenia, or functional asplenia;
    * Have a history of myocarditis, pericarditis or idiopathic cardiomyopathy, or have any disease that increases the risk of myocarditis or pericarditis;
    * Has a history of inflammatory demyelinating neurological disorders such as Guillain-Barré syndrome;
    * Has severe or unstable cardiovascular diseases, diabetes, diseases of the blood and lymphatic systems, immune system diseases, liver and kidney diseases, respiratory diseases, metabolic and skeletal diseases, or malignant tumors;
    * Has contraindications for intramuscular injections and blood drawing;
11. Have a history of major surgery within 3 months prior to randomization or planned surgery during the trial.
12. Drug/alcohol abuse within 1 year prior to randomization, deemed by investigators to impact safety assessment or compliance.
13. Have received lipid nanoparticle (LNP)-based vaccines/medications within 1 year prior to randomization; current participation in other RSV-related trials; OR planned to participate in other clinical trials during this study.
14. The investigators evaluated that any disease or condition of the participants might place them at an unacceptable risk; The participants failed to meet the requirements of the protocol; circumstances that interfered with the assessment of the vaccine response.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Solicited Local and Systemic Adverse Reactions Through 14 Days After Initial Vaccination | From initial vaccination up to14 days post initial vaccination
Percentage of Participants With Unsolicited Adverse Events (AEs) Through 28 Days After Initial Vaccination | From initial vaccination up to 28 days post initial vaccination
Percentage of Participants With Unsolicited AEs Through 30 Minutes After Initial Vaccination | From initial vaccination up to 30 minutes post initial vaccination
Percentage of Participants With Any Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) During Study | Through study completion, about 3 years at most
Percentage of Abnormal Results of Hematology On Day 3 After Initial Vaccination Compared with Baseline | From initial vaccination up to 3 days post initial vaccination
Percentage of Abnormal Results of Clinical Chemistry On Day 3 After Initial Vaccination Compared with Baseline | From initial vaccination up to 3 days post initial vaccination
Percentage of Abnormal Results of Coagulation On Day 3 After Initial Vaccination Compared with Baseline | From initial vaccination up to 3 days post initial vaccination
Percentage of Participants With Any AEs Leading to Discontinuation of Vaccination or Withdrawal From The Study | Through study completion, about 3 years at most
Geometric mean concentration (GMC) for Pre-F Specific IgG Antibody Against RSV A and RSV B | 1 month post-initial vaccination
Geometric Mean Fold Rise (GMFR) for Pre-F Specific IgG Antibody Against RSV A and RSV B | 1 month post-initial vaccination
Seroconversion Rate (SCR) for Pre-F Specific IgG Antibody Against RSV A and RSV B | 1 month post-initial vaccination
Geometric mean titer (GMT) for Neutralizing Antibody Against RSV A and RSV B | 1 month post-initial vaccination
GMFR for Neutralizing Antibody Against RSV A and RSV B | 1 month post-initial vaccination
SCR for Neutralizing Antibody Against RSV A and RSV B | 1 month post-initial vaccination

SECONDARY OUTCOMES:
GMC for Pre-F Specific IgG Antibody Against RSV A and RSV B | 3, 6 and 12 months post-initial vaccination
GMFR for Pre-F Specific IgG Antibody Against RSV A and RSV B | 3, 6 and 12 months post-initial vaccination
SCR for Pre-F Specific IgG Antibody Against RSV A and RSV B | 3, 6 and 12 months post-initial vaccination
GMT for Neutralizing Antibody Against RSV A and RSV B | 3, 6 and 12 months post-initial vaccination
GMFR for Neutralizing Antibody Against RSV A and RSV B | 3, 6 and 12 months post-initial vaccination
SCR for Neutralizing Antibody Against RSV A and RSV B | 3, 6 and 12 months post-initial vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided